CLINICAL TRIAL: NCT05557799
Title: Photobiomodulation in Post Menopause Genitourinary Syndrome - Study Protocol for a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Photobiomodulation in Post Menopause Genitourinary Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGPM
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Postmenopausal Symptoms
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the participant nor the outcome assessor will know to which group the participant belongs, seeing as laser application will be simulated in the placebo group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation group (Active Comparator): Participants in this group will receive photobiomodulation with a vaginal diode laser and its introit.
  Interventions: Radiation: Photobiomodulation
- Placebo group (Placebo Comparator): Participants in this group will receive simulated photobiomodulation, with the laser device turned off.
  Interventions: Radiation: Placebo Photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — The treatment group will receive four consecutive applications, using laser diode DMC (808 nm), 4J per point, 100mW of power, 510mW/cm², beam area of 0.2cm², 8 sites in the external vagina, for 40s in each site, once per week for 4 weeks.
  Arms: Photobiomodulation group
Radiation: Placebo Photobiomodulation — The Placebo Group will receive the same four consecutive applications, but with the laser turned off.
  Arms: Placebo group

SUMMARY:
The goal of this project is to evaluate the clinical response of patients with symptoms of genitourinary menopause syndrome after the application of photobiomodulation in the vagina and its introit. METHOD: In this randomized, double-blind, placebo-controlled study protocol, women over 50 years of age who are in the postmenopausal period (amenorrhea for at least 12 months, with no pathology involved) with one or more symptoms of PGS will be selected. Participants included in the study will be randomly divided into two groups: group A, which will receive photobiomodulation with a vaginal diode laser and its introit and group B (placebo) with the laser device turned off. Both treatments will be maintained for 4 consecutive weeks.The treatment group (n=30) will receive four consecutive applications, using laser diode DMC (808 nm), 4J per point, 100mW of power, 510mW/cm², beam area of 0.2cm², 8 sites in the external vagina, for the 40s in each site, once per week for 4 weeks. The Placebo Group (n=30) will be handled as treated, but with the laser turned off. Quality of life will be analyzed using the female sexual functioning index (FSFI-6), the urinary incontinence questionnaire (ICIQ-SF), the intensity of menopausal symptoms will be evaluated using a visual analogue scale (VAS), the vulvo vaginal atrophy will be measured by the Vaginal Health Index (VHI) and compared between groups. Also, the vaginal temperature will be measured using a thermal camera, as well as the pressure of the pelvic floor force (vaginal dynamometer) and a 1-hour Pad Test will be performed to quantify the urinary loss. The data will be tested for normality using the Shapiro Wilks test and, if they present a parametric distribution, they will be represented by means of their respective means and standard deviations.

ELIGIBILITY:
Inclusion Criteria:

* Women over 50 years of age who are in the postmenopausal period (amenorrhea for at least 12 months, with no pathology involved);
* With one or more symptoms of UGS (dyspareunia, dryness, irritation and vaginal burning and/or discomfort, vaginal atrophy, vaginal and vulvar dryness, dysuria, frequency, recurrent urinary infections);
* With complaints of stress and/or urge urinary incontinence;
* Who have cervical cytopathology (Pap smear) within the normal range performed in the last year and are not in use of hormonal medication to treat menopausal symptoms in the last 6 months.

Exclusion Criteria:

* Participants with explicit refusal of the patient to participate in the researc;
* History of bilateral oophorectomy and diseases such as: recent AMI (Acute Myocardial Infarction), neoplasms, history of thrombosis, liver failure, uncontrolled genital bleeding, genital condylomatosis, active genital herpes, lower genital tract surgeries that make treatment impossible.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the Female Sexual Function Index (FSFI) | Baseline and the 4 weeks of treatment.
  The FSFI or female sexual function index is a specific and multidimensional questionnaire to assess female sexual response, accessing 6 domains: desire, arousal, lubrication, orgasm, satisfaction and pain evaluated in 19 questions about sexual activity in the last 4 weeks. In order to obtain the total score of the scale, the scores for each domain are added up, and for higher scores, better sexual function is considered, and the threshold for sexual dysfunction is a score of 2678. Based on the value of the total score, it would be possible discriminate between populations at higher and lower risk of experiencing sexual dysfunction.

SECONDARY OUTCOMES:
Changes in the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) | Baseline and the 4 weeks of treatment.
  This questionnaire has a score from zero to 21 points, with zero indicating the absence of symptoms and the greater the sum of the points, the greater the impact and severity of urinary incontinence (UI) symptoms. The maximum sum of the response values indicates a score of 21 points, referring to a high impact of UI on the individual's life.
Changes in the Vaginal Health Index Score | Baseline and the 4 weeks of treatment.
  It consists of a clinical analysis during the speculum examination of 5 parameters: elasticity, pH, mucosal appearance, humidity and the presence of vaginal secretion. Each aspect evaluated receives a score, which varies from 1 to 5. The score may vary from 5 to 25, and a diagnosis of Vulvo Vaginal Atrophy (VVA) is considered when the values are less than or equal to 15, the maximum score of 25 points means absence of clinical signs of vulvovaginal atrophy. This assessment will be performed by a qualified professional during the physical examination.
Changes in the Vaginal pH | Baseline and the 4 weeks of treatment.
  The evaluation of the vaginal pH will be carried out through a pH indicator strip, which when inserted in the middle third of the vagina in contact with the mucosa, has the color of the strip changed. Measurement of the vaginal cul-de-sac is avoided, because contact with mucus, blood or semen can alter the reading. The nitrazine tape must remain in contact with the vaginal wall for 5 seconds for later checking the pH on the colorimetric scale provided by the manufacturer. Normal vaginal pH is acidic, during menacme, it should be maintained between 3.8 and 4.5.
Changes in Pain using a Visual Analog Scale (VAS) | Baseline and the 4 weeks of treatment.
  A VAS will be used to evaluate the vaginal complaints of the participants. They will receive a figure of a ruler with marks from 0 to 10, whose one end indicates complete absence of symptoms and the other indicates the worst possible symptom. For analysis of the Visual and Analog Scale of Symptoms of Genitourinary Syndrome (GUS) (VAS - SGU), the sum of one to twelve points will classify the symptoms from mild to severe.
Changes in the Pelvic Floor Muscles (PFMs) | Baseline and once a week for 4 weeks
  The pressure sensor (dynamometer) will be introduced into the vaginal canal, and the resting vaginal pressure (resting muscles) will be quantified. The device will be calibrated, zeroed and it will be asked for the participant to contract their PFMs inwards and upwards as hard as possible 3 times and maintain the contraction for at least five seconds (maximum vaginal pressure), with an interval of 30 seconds between each pull.
Changes in Urinary Loss using Ped-Test | Baseline, the 4 weeks of treatment and 90 days after treatment.
  The procedure for performing the Ped-test will be as follows: initially, the participant will be asked to place an absorbent with a previously measured weight close to the external urethral meatus. Then, she will be given a 500 mL bottle of water to drink and wait for 15 minutes. Afterwards, the participant will be asked to perform some actions simulating activities of daily living. After carrying out the proposed activities, the absorbent will be removed and weighed on a precision scale, with a minimum reading of 0.1 mg and a maximum capacity of 220 g. Urinary losses are evaluated and classified as follows: losses of up to 1 g are considered insignificant; between 1.1 and 9.9 g are classified as light losses; between 10 and 49.9 g are moderate losses; and above 50 g, severe losses.
Changes in Vulva Temperature | Baseline and and once a week for 4 weeks
  The temperature of the vulva, in Celsius degrees, will be evaluated at the eight points of radiation in the vulvar region, with a digital infrared thermometer, which will allow measurement without physical contact. The average of the eight readings will be calculated before and after the diode laser procedure in the 4 consecutive weekly sessions.

REFERENCES:
- [Derived] Pereira SRDS, Mesquita-Ferrari RA, Salviatto LTC, Bezerra CDDS, Dalapria V, Mello EDS, Almeida-Lopes L, Bossini PS, Goncalves MLL, Deana AM. Photobiomodulation in post menopause genitourinary syndrome-Study protocol for a randomized, double-blind, controlled clinical protocol. PLoS One. 2024 Dec 2;19(12):e0313324. doi: 10.1371/journal.pone.0313324. eCollection 2024. PMID 39621728